CLINICAL TRIAL: NCT04873141
Title: Tocilizumab and Cytokine Release Syndrome (CRS) In Covid-19 Pneumonia: Experience From Single Center of Pakistan
Brief Title: Tocilizumab and Cytokine Release Syndrome (CRS) In Covid-19 Pneumonia
Status: Completed | Type: Observational
Sponsor: Shaheed Zulfiqar Ali Bhutto Medical University (Other)
Responsible Party: Principal Investigator, Fibhaa Syed, Assistant Professor, Shaheed Zulfiqar Ali Bhutto Medical University
Other Study IDs: Tocilizumab and CRS
Record Dates: First submitted 2021-04-28; First posted 2021-05-05 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-05

CONDITIONS: Cytokine Release Syndrome; Covid-19 Pneumonia
Keywords: Cytokine Release Syndrome; Covid-19 Pneumonia; Tocilizumab
MeSH Terms: conditions — Cytokine Release Syndrome | interventions — tocilizumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Case Group: All the patients suffering from severe covid pneumonia and laboratory parameter suggestive of cytokine release syndrome.
  Interventions: Drug: Tocilizumab 200 Mg/10 mL (20 Mg/mL) INTRAVEN VIAL (ML)

INTERVENTIONS:
Drug: Tocilizumab 200 Mg/10 mL (20 Mg/mL) INTRAVEN VIAL (ML) — Tocilizumab was given according to weight in patients with cytokinme releasew syndrome (CRS).
  Other Names: Actemra

SUMMARY:
Tocilizumab (TCZ), interleukin-6 (IL-6), newly appeared as treatment of cytokine release syndrome (CRS) in patients with severe covid-19 associated pneumonia. In the present study, we aimed to discuss the treatment response of TCZ therapy in COVID-19 infected patients.

DETAILED DESCRIPTION:
This observational study was designed just to visualize the efficacy and safety of Tocilizumab, an antibody anti-IL-6 receptor in patients with moderate to severe COVID-19 with increased inflammatory markers.Patients will be followed until Day 29 after randomization.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old; Clinical diagnosis of SARS-CoV-2 virus by PCR, or by other approved diagnostic methodology, or, with presumptive diagnosis of COVID-19 (other respiratory causes ruled out and COVID-19 test pending); Hospitalized with COVID-19-induced pneumonia; Elevated CRP, D-Dimers or ferritin levels; Bodyweight ≥ 40kg.

Exclusion Criteria:

* Eligible patients must not have a history of hypersensitivity to any drugs or metabolites of similar chemical classes as canakinumab; Use of tocilizumab within 3 weeks prior; Suspected or known active bacterial, fungal, or parasitic infection (besides COVID-19); Patients with significant neutropenia (ANC <1000/mm3); Treatment with an investigational drug within 5 half-lives or 30 days (whichever is longer) prior to tocilizumab dose.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of age (18-all) and suffering from COVID- 19 severe pneumonia
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2020-04-28 (Actual); Primary Completion 2020-06-22 (Actual); Study Completion 2020-06-22 (Actual)

PRIMARY OUTCOMES:
Mortality Rate | 28 days
  Patient admitted with cytokine release syndrome and given Tocilizumab and primary outcome was death within hospital.
Time to discharge | 28 days
  Time to Hospital Discharge or "Ready for Discharge" as evidenced by normal body temperature and respiratory rate, and stable oxygen saturation on ambient air or >/= 2 liters (L) supplemental oxygen.

SECONDARY OUTCOMES:
Laboratory parameters | 30 days
  All the specialized labs (Serum Ferritin, CRP, D- Dimer . IL-6) will be observed till its normal level.
Oxygen Saturation | 30 days
  Patients who were given Tocilizumab, observed for demand of oxygen therapy to see decremental response of oxygen, whether its decreasing or increasing after tocilizumab dosing and it will be observed both in pulse oximeter and oxygen given in L/min.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Hassan, MD, Principal Investigator — Shaheed Zulfiqar Ali Bhutto Medical University
Locations (1):
- Shaheed Zulfiqar Ali Bhutto Medical University, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No
The study was completed and we retrospectively putting data of a prospective study.